CLINICAL TRIAL: NCT05856110
Title: Coronary Computed Tomography Angiography and Functional Analysis in Risk Stratification of Coronary Artery Disease: A Prospective, Multi-center Cohort Study
Brief Title: Risk Evaluation by COronary CTA and Artificial IntelliGence Based fuNctIonal analyZing tEchniques - II
Acronym: RECOGNIZE-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, Director of Cardiology, Director of cardiovascular catherization lab, Principle Investigator, Ruijin Hospital
Other Study IDs: 2022YFC2533502-2
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary CTA; CT-FFR; Risk Stratification; Artificial Intelligence
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter, prospective clinical cohort study. The study intends to continuously enroll patients with coronary heart disease. All subjects will undergo coronary CTA (followed by anatomic, functional and radiomics analysis), proteomics research as well as clinical follow-up of cardiovascular events. The purpose of this study is to establish a new, non-invasive cardiovascular disease risk stratification system.

DETAILED DESCRIPTION:
Coronary angiography has been the gold standard for the diagnosis of coronary heart disease and PCI decision-making. However, the value of CAG in risk stratification is limited due to its invasive nature and lack of ability to evaluate coronary physiology and plaque characteristics, which often leads to over-treatment or under-treatment. In recent years, with the development and improvement of imaging technology, the resolution and diagnostic accuracy of coronary artery CTA have been greatly improved, and the subsequent anatomy and function (non-invasive CT-FFR, etc.) have made the assessment of coronary artery lesion risk multi-dimensional. Comprehensive and accurate coronary artery CTA scan plays a positive role in establishing the appropriate standard for PCI and improving the prognosis of patients. However, the existing problems of coronary artery CTA are insufficient imaging studies, complex image analysis, inconsistent diagnostic criteria, and insufficient clinical evidence. This study is one of the series of clinical studies on the topic of "Risk Evaluation by COronary Computed Tomography and Artificial Intelligence Based fuNctIonal analyZing tEchniques (RECOGNIZE)". The purpose of the study is to evaluate the accuracy of early identification of cardiovascular high-risk groups based on the functional evaluation model based on coronary CTA images through a multi-center, prospective clinical cohort study, so as to establish an early, non-invasive and accurate risk classification of cardiovascular events in coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Clinically significant angina pectoris, suspecting coronary artery disease

Exclusion Criteria:

* Unsuitable for coronary CTA (such as severe renal impairment, uncontrolled thyroid condition, allergic to iodine, etc.)
* Without a visible plaque (defined as ≥ 30% stenosis) in major coronary arteries in coronary CTA
* Prior history of myocardial infarction or heart failure
* Prior history of percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
* Severe renal or liver failure
* Familial hypercholesterolemia
* Estimated survival ≤1 year
* Malignant tumor
* Poor coordinance, unable to follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a multi-center cohort study. Patients with clinical angina pectoris and suspected coronary artery disease from nine clinical centers across P.R. China, including outpatient and hospitalized patients, are consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 2 years
  Including cardiovascular death, myocardial infarction, and stroke

SECONDARY OUTCOMES:
Cardiovascular death | 2 years
  Death due to cardiovascular events
Myocardial infarction | 2 years
  Including STEMI and NSTEMI
Stroke | 2 years
  Including ischemic and hemorrhagic stroke
Coronary Revascularization | 2 years
  Including percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG)

CONTACTS AND LOCATIONS:
Overall Officials: Ruiyan Zhang, M.D., Ph.D., Principal Investigator — Ruijin Hospital; Lin Lu, M.D., Study Chair — Ruijin Hospital; Fei Ye, M.D., Study Chair — First Hospital of Nanjing; Yachen Zhang, M.D., Study Chair — Xinhua Hospital, Shanghai Jiaotong University School of Medicine; Tian Xie, M.D., Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Lei Liu, M.D., Study Chair — First Affiliated Hospital of Harbin Medical University; Xiaolei Yang, M.D., Study Chair — The First Affiliated Hospital of Dalian Medical University; Run Guo, M.D., Study Chair — Cangzhou Center Hospital; Yingying Guo, M.D., Study Chair — The First Affiliated Hospital of Zhengzhou University; Geng Wang, M.D., Study Chair — The General Hospital of Northern Theater Command
Locations (9):
- China (9):
  - Cangzhou Center Hospital, Cangzhou, Hebei
  - First affiliated hospital of Harbin Medical University, Harbin, Heilongjiang
  - First affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Techonology, Wuhan, Hubei
  - First Hospital of Nanjing, Nanjing, Jiangsu
  - First affiliated hospital of Dalian Medical College, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided